CLINICAL TRIAL: NCT06257433
Title: The Influence of Mesolimbic-hippocampal Interactions on Episodic Memory During Active Information Seeking
Brief Title: InformationSeekingMesolimbicEngagementStudy2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01DA055259-2; R01DA055259 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Motivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Motivation (Experimental): Trials in which participants are motivated by hypothesis testing or not.
  Interventions: Behavioral: Task Instructions

INTERVENTIONS:
Behavioral: Task Instructions — Participants will be given cued instructions as to whether they are in a high or low motivation condition

SUMMARY:
Participants will complete a treasure task during neuroimaging where they have to learn which keys open a treasure chest, and then they are tested on the contents of the treasure chest.

DETAILED DESCRIPTION:
Study 2 will use a treasure task (employed in C.2.1.1), in which participants select amongst 3 keys to learn which feature of keys unlocks the treasure chest, revealing a trial unique object image (Fig. 8b). On each encoding trial participants view three multi-featural keys and a treasure chest. Each key varies on three dimensions: color (red, blue, yellow), shape of the handle (square, circle, triangle), and number of ridges (one, two, three). On each trial, all 9 dimensions of the keys are represented, but the dimensions represented on each key are randomized across trials. During hypothesis testing runs, participants are instructed to find the feature of a key that opens the treasure chest to reveal a trial-unique image. Critically, there is one target feature of a key that deterministically opens the treasure chest. The target feature of the key randomly changes after participants successfully open the chest 4 consecutive times. This design manipulates goal-oriented exploration by allowing participants to resolve uncertainty until they identify the target feature of the key. Uncertainty resolution is the greatest after the target features switches and incrementally reduces via individuals' active hypothesis testing. During control runs, participants will be instructed to select specific keys, and key selection and outcomes will be yolked to prior hypothesis testing runs. Participants will complete 3 runs of hypothesis testing runs and 3 control runs. Trial number for each run is determined by participant behavior, in that hypothesis testing runs end when participants complete 4 rule switches (~30 trials). Encoding is incidental in this task. Following encoding, participants will complete an immediate and delayed item memory test. On each trial, participants will view objects from the hypothesis testing and control conditions as well as new foil objects. Memory will be tested for half the stimuli immediately and at a 24-hour delay. These memory measures will be related to uncertainty resolution estimated by reinforcement learning, to determine how prior knowledge during information seeking has subsequent effects on memory.

ELIGIBILITY:
Inclusion Criteria:

* 20/40 far acuity (either corrected or uncorrected)
* In good medical health

Exclusion Criteria:

* History of head injury
* History of illness with Central Nervous Systems implications
* On Medications that Affect blood flow response and alertness
* Consumption of smoking and/or coffee 30 minutes prior to laboratory testing
* Placement of a device contraindicated for magnetic resonance imaging including cardia pacemaker, aneurysm clip, cochlear implants, pregnancy, intra-uterine device, shrapnel, metal fragments in the eyes, neurostimulators
* Weight > 250lbs
* Claustrophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Mesolimbic Hippocampal Interactions | During Procedure
  Functional Magnetic Resonance Imaging Activation characterizing Mesolimbic-Hippocampal Interactions
Episodic Memory | 24-hours After Procedure
  Item and Associative Memory for memoranda shown during the task

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared on the open science framework.
Supporting Information: Analytic Code
Time Frame: Data will be shared within 1 year of study completion, and it will be available for at least 10 years.